CLINICAL TRIAL: NCT07297576
Title: Safety and Feasibility of Sulforaphane to Promote Early Haematopoietic Recovery After Cord Blood Transplantation A Single-arm, Open, Single-centre Clinical Study
Brief Title: Safety and Feasibility of Sulforaphane to Promote Early Haematopoietic Recovery After Cord Blood Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025085
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-09

CONDITIONS: ALL (Acute B-Lymphoblastic Leukemia); AML (Acute Myelogenous Leukemia; MDS (Myelodysplastic Syndrome)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — sulforaphane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Test group (Experimental): For the Aspirin arm, 30mg/tablet of the antioxidant substance radicicolothionein for oral administration, two tablets each time, three times a day; unrelated umbilical cord
  Interventions: Dietary Supplement: Sulforaphane

INTERVENTIONS:
Dietary Supplement: Sulforaphane — For the Aspirin arm, 30mg/tablet of the antioxidant substance radicicolothionein for oral administration, 2 tablets each time, three times a day; unrelated umbilical cord

SUMMARY:
Umbilical cord blood (UCB) is rich in haematopoietic stem progenitor cells and immune cells, and is used for transplantation for a variety of haematological disorders with the advantages of low mating requirements and fewer transplant complications. By March 2025 China's seven (eight) public cord blood stem cell banks had frozen more than 280,000 public umbilical cord blood, while the percentage of those frozen for ≥10 years was 26%, making clinical application a concern. The previous study showed that long-term freezing impairs cellular mitochondrial function leading to decreased reconstruction of cord blood haematopoietic stem progenitor cells and impaired differentiation into the megakaryotic lineage, and that intervention with the antioxidant radicicol thiols (SFN) can partially rescue the cellular functional damage caused by freezing. The findings were based on immunodeficient animals, and clinical studies are urgently needed to determine whether SFN intervention can promote post-transplant haematopoietic reconstitution in patients with long term cryopreserved (≥10 years) UCB. In this project, the investigators propose to conduct a single-arm, open, single-centre phase I-II clinical study on the safety and feasibility of dietary supplement SFN to promote early haematopoietic restoration after cord blood transplantation to evaluate the safety and feasibility of the use of long-frozen UCB for peri-infusion SFN use in adult transplant recipients, and to reveal the effect of peri-infusion SFN use on neutrophil implantation. This project will provide scientific guidance to promote the clinical application of long-term cryopreserved UCB, as well as key data to optimise the clinical transplantation strategy of UCB and expand its application.

DETAILED DESCRIPTION:
Please see the detailed description in following content

ELIGIBILITY:
Inclusion criteria：

1. Patients with high-risk haematological malignancies: including AML, ALL, high-risk MDS
2. Age: ≥18 years
3. Karnofsky score ≥70%, Eastern Cooperative Oncology Group (ECOG) physical status ≤2 points
4. Selection of non-haematopoietic cord blood: donor-recipient HLA high-resolution compatibility ≥4/6, 7/10 and CD34 cells ≥0.83×105/kg (recipient's body weight), meeting the above criteria, only cord blood with a freezing time of ≥10 years can be found in China's public umbilical cord blood stem cell banks.

Exclusion criteria：

1. Patients who test positive for the following pathogens: HIV (HIV-1/2), human cytomegalovirus (HCMV-DNA), EBV (EBV-DNA), Hepatitis B (positive for Hepatitis B Surface Antigen (HBsAg) or Hepatitis B DNA (HBV-DNA)), Hepatitis C Antibody (HCV-Ab), Treponema pallidum Antibody (TP-Ab).
2. Active bacterial, viral, fungal or parasitic infections of clinical significance as judged by the investigator at the time of screening
3. Willing donors with full HLA compatibility and eligible for allogeneic haematopoietic stem cell transplantation
4. Previous gene therapy or allogeneic haematopoietic stem cell transplant recipients
5. Immediate family members with known or suspected familial cancer syndromes (including but not limited to hereditary breast and ovarian cancer syndromes, hereditary non-polyposis colorectal cancer syndromes, familial adenomatous polyposis, etc.)
6. Confirmed diagnosis of a major mental illness or predisposition to mental illness that would seriously affect the ability to participate in clinical research
7. History of major organ injury, including: Liver lesions: liver function tests suggesting AST or ALT > 3 × ULN; total serum bilirubin > 2.5 × ULN; total bilirubin > 3 × ULN and direct bilirubin > 2.5 × ULN if consistent with Gilbert's syndrome; history of hepatic pontine fibrosis, cirrhosis, and the presence of active hepatitis; Cardiac lesions: left ventricular ejection fraction ("LVEF") < 45%; New York Heart Association (NYHA) class III or IV congestive heart failure (see Appendix 1 for classifications of heart failure); severe heart failure requiring treatment. Cardiac pathology: left ventricular ejection fraction (LVEF) <45%; New York Heart Association (NYHA) class III or IV congestive heart failure (see Appendix 1 for NYHA heart failure classification); severe arrhythmia requiring treatment; uncontrolled hypertension or unstable angina; myocardial infarction or bypass or stent surgery within 12 months prior to enrolment; clinically significant valvular disease; calculated eGFR <60mL/min/1.73m2 and direct bilirubin >1.73m2; history of hepatic bridging fibrosis and cirrhosis; and presence of active hepatitis. Lung function: FEV1/FVC <60% and/or diffusion function <60% of predicted value; clinically significant evidence of pulmonary hypertension requiring medical intervention.
8. Uncorrectable coagulation disorders or history of severe bleeding disorders
9. Any other condition that, in the opinion of the doctor, makes the subject unsuitable for haematopoietic stem cell transplantation
10. Known allergy to the test drug or ingredients
11. Have participated or are participating in other interventional clinical studies within 3 months prior to screening
12. Live vaccination within 6 weeks prior to screening
13. Pregnant or breastfeeding women
14. Subjects did not follow the study protocol well
15. Any other condition deemed by the investigator to be unsuitable for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of the occurrence of adverse events, including non-haematological adverse events of grade 3 or higher | 2 months post-transplant
  Based on CTCAE (Common Terminology Criteria for Adverse Events) grading, determine the need for dose reduction or suspension of medication; observe the incidence of transplant-related complications acute GVHD, the incidence of infections, the transplant-related mortality Rate (TRM)
Time to neutrophil recovery after UCBT | 3 months post-transplant
  Blood routine test

CONTACTS AND LOCATIONS:
Overall Officials: Fang Dong, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, Tianjin, China
Locations (1):
- Institute of Hematology, Blood Diseases Hospital, Tianjing, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT07297576/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT07297576/ICF_001.pdf